CLINICAL TRIAL: NCT02865278
Title: Evaluation of the Bioavailability of Polyphenols From a Red Grape Extract-based Drink and the Acute Effects of Its Consumption on Glucose and Lipid Response During the Subsequent Meal
Brief Title: Bioavailability of the Polyphenols Contained in a Red Grape Extract-based Drink and Their Metabolic Effects
Acronym: BIOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, rivellese angela, Full professor, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 29/16
Record Dates: First submitted 2016-07-15; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polyphenol-rich drink (Experimental): The participants consume the polyphenol-rich drink. After 3 hours they consume a standard meal to evaluate whether the metabolic response may be influenced by polyphenols.
  Interventions: Other: Standard meal
- Placebo drink (Placebo Comparator): The participants consume the control drink.After 3 hours they consume a standard meal to evaluate the metabolic response after a placebo.
  Interventions: Other: Standard meal

INTERVENTIONS:
Other: Standard meal — The participants consume the drink, experimental or placebo drink. After 3 hours they consume a standard meal (905 kcal, 15% protein, 46% fat, 39% CHO). Blood samples are taken at fasting, over 3 hours after drink consumption and over 5 hours after the test meal to evaluate metabolic response. Fasting and 48h-urine are collected to evaluate bioavailability of polyphenol.

SUMMARY:
Randomized placebo-controlled crossover study during which participants undergo two different experimental days. The participants consume a red grape based- drink (polyphenols: 300 mg/100 ml and sugar: 9.8g/100 ml) or a placebo (no polyphenols and sugar: 9.8g/100 ml). After 3 hours they consume a test meal (905 kcal, 15% protein, 46% fat, 39% CHO). Blood samples are taken at fasting, over 3 hours after drink consumption and over 5 hours after the test meal to evaluate metabolic response. Fasting and 48h-urine are collected to evaluate bioavailability.

ELIGIBILITY:
Inclusion Criteria:

* BMI >25 and <35 kg/m2
* Total cholesterol <250 mg/dl
* Triglyceride < 200 mg/dl.
* Fasting glucose <100 mg/dl

Exclusion Criteria:

* Cardiovascular events (IMA or stroke) in the 6 months prior to the study
* Kidney or liver failure
* Anemia (Hb <12 g/dl)
* Any chronic disease
* Intense physical activity
* Dietary supplements

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Phenolic metabolites in urine | 48 hours
  GCxGC-MS

SECONDARY OUTCOMES:
Glucose response | 8 hours
  Enzymatic colorimetric methods
Inflammation | 8 hours
  Multiplex Detection Immunoassays
Oxidative stress (urinary isoprostanes) | 8 hours
  EIA
Triglyceride response | 8 hours
  Enzymatic colorimetric methods

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Costabile G, Vitale M, Luongo D, Naviglio D, Vetrani C, Ciciola P, Tura A, Castello F, Mena P, Del Rio D, Capaldo B, Rivellese AA, Riccardi G, Giacco R. Grape pomace polyphenols improve insulin response to a standard meal in healthy individuals: A pilot study. Clin Nutr. 2019 Dec;38(6):2727-2734. doi: 10.1016/j.clnu.2018.11.028. Epub 2018 Dec 7. PMID 30573355